CLINICAL TRIAL: NCT07237594
Title: A Feasibility Study Utilizing IL-17 Blockade to Decrease Risk of Immune Related Adverse Events
Brief Title: IL-17 Blockade to Decrease irAEs (REPLAY)
Acronym: REPLAY
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00118701
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Secukinumab (Experimental): Participants will first undergo pre-treatment with secukinumab (300mg subcutaneously) within 1 to 7 days prior to resumption of ICI treatment. Participants will then undergo anti-PD-1 therapy, anti PD-1 plus anti LAG3 (relatlimab) or anti-PD-1 plus anti CTLA-4 therapy at the discretion of their treating physician. Participants will concurrently receive secukinumab 300mg subcutaneously weekly for the first 4 weeks of treatment and then every 4 weeks.
  Interventions: Drug: Secukinumab Injection

INTERVENTIONS:
Drug: Secukinumab Injection — Secukinumab 300mg subcutaneously

SUMMARY:
The primary objective of this study is to determine the safety and feasibility of administering an IL-17A (human IgG1κ) monoclonal antibody, (Secukinumab, Cosentyx®) to participants with metastatic melanoma who have previously received immune checkpoint inhibitor (ICI) therapy, experienced an immune related adverse event (colitis, hepatitis, skin rash, psoriatic arthritis) to ICI, and are re-initiating ICI therapy.

DETAILED DESCRIPTION:
Participants will receive pre-treatment (pre-ICI) with secukinumab (300mg) within 1 to 7 days prior to the initial ICI dose. Participants will then resume ICI therapy (the specific ICI agent and dose are determined by the treating physician per their standard practice). Participants will receive secukinumab weekly for the first 4 weeks, and then once every 4 weeks thereafter until grade 3 side effect occurs or ICI is discontinued.

Participants will have AE (adverse event) assessments at each study visit. Disease assessments via CT scans will be performed every 12 weeks with iRECIST/RECIST. Research blood samples and tumor tissue will be collected. All participants will be followed by phone call or medical record review for survival for up to three years. Participants who come off for reasons other than disease progression will also be followed with CT scans every 12 weeks until progression for up to two years.

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed advanced metastatic melanoma
2. Participants of any gender who are at least 18 years of age on the day of signing informed consent
3. Participants must be planned or scheduled by their treating physician to receive PD-1 therapy or PD-1 plus anti LAG3 or PD-1 plus anti CTLA-4 therapy as standard of care. Patients should either be restarting the same ICI regimen which contributed to the prior toxicity or have a clinical need to escalate to doublet (combination) ICI therapy, plan for therapy should be reviewed by the PI of this study.
4. Participant (or legally acceptable representative if applicable) provides written informed consent for the trial
5. Participant must have had prior treatment with ICI therapy (either PD-1 therapy or PD-1 plus anti LAG3 or PD-1 plus anti CTLA-4 therapy as standard of care) and experienced grade 2 or higher immune-related colitis, hepatitis, or skin rash leading to treatment interruption or discontinuation or requiring steroid administration (systemic or topical).

   * Note that patients who experience more than one irAEs are eligible to participate
6. Adequate organ function as defined below. Standard of care labs drawn within 42 days prior to consent may be used for the purposes of determining eligibility.

   * Absolute Neutrophil Count (ANC) ≥ 1500/µL
   * Platelets ≥ 100,000/µL
   * Hemoglobin* ≥ 9.0 g/dL or ≥ 5.6 mmol/L *Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within the previous 2 weeks
   * AST/ALT 2.5x upper limit of normal

Exclusion Criteria:

1. Uveal melanoma
2. Any participants known to be pregnant or breastfeeding.
3. Known diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone or equivalent), or any other form of immunosuppressive therapy within 7 days prior to first research biopsy
4. Patients with symptomatic CNS metastases and/or carcinomatous meningitis

   * Patients with asymptomatic, clinically stable CNS metastases are allowed provided they do not require steroid treatment
5. History of or active (non-infectious) pneumonitis that required steroids
6. Active infection requiring systemic therapy
7. Known history of Human Immunodeficiency Virus (HIV) infection
8. Known history of Hepatitis B or known active Hepatitis C virus infection. NOTE: no testing for Hepatitis B or Hepatitis C is required
9. Known history of active TB (Bacillus Tuberculosis)
10. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with subject's participation for the full duration of the study, or make it not in the best interest of the subject to participate, in the opinion of the treating physician
11. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
12. History of allogenic tissue or solid organ transplant
13. History of active autoimmune disease requiring systemic therapy within the past 12 months, with the exception of ICI induced irAEs.
14. Has not been treated with secukinumab within the last 12 months
15. History of prior cardiac, neurologic, ocular IRAE related to ICI; history of blistering cutaneous IRAE related to ICI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of administering an IL-17A (human IgG1κ) monoclonal antibody (secukinumab) as determined by occurrence of immune-related Adverse Events (irAEs) | Until grade 3 side effect occurs or three years, whichever comes first
  Participants will be assessed for AEs at each study visit. AEs are graded by NCI-CTCAE v5.0 criteria.
Feasibility of administering an IL-17A (human IgG1κ) monoclonal antibody (secukinumab) as determined by occurrence of immune-related Adverse Events (irAEs) | Until grade 3 side effect occurs or three years, whichever comes first
  Participants will be assessed for AEs at each study visit. AEs are graded by NCI-CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: April Salama, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No